CLINICAL TRIAL: NCT03121716
Title: An Open-Label, Single Center, Nonrandomized, Phase 1 Study to Evaluate Safety and Efficacy of Using the Combination Treatment of SHR-1210, Gemcitabine and Cis-platinum by Recurrent and Metastatic NPC
Brief Title: A Study to Evaluate the Safety and Efficacy of SHR-1210, Gemcitabine and Cis-platinum by R/M NPC Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHR-1210-104
Record Dates: First submitted 2017-04-13; First posted 2017-04-20 (Actual); Last update posted 2022-07-12 (Actual); Status verified 2018-12

CONDITIONS: Nasopharyngeal Carcinoma
MeSH Terms: conditions — Nasopharyngeal Carcinoma | interventions — camrelizumab; Gemcitabine; Injections; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SHR-1210, gemcitabine and cis-platinum (Experimental): Subjects receive SHR-1210 200mg (Day 1) and gemcitabine 1000mg/m2 (Day 1 and Day 8)and cis-platinum 80mg/m2 (Day 1) of each 21-day cycle for at most 6 cycles, followed by SHR-1210 200mg every three weeks (Q3W) maintenance for the remainder of the study or until documented PD.
  Interventions: Biological: SHR-1210; Drug: Gemcitabine; Drug: cis-platinum

INTERVENTIONS:
Biological: SHR-1210 — SHR-1210 is a humanized anti-PD1 IgG4 monoclonal antibody.
Drug: Gemcitabine — gemcitabine
  Other Names: Gemcitabine Hydrochloride for Injection
Drug: cis-platinum — cis-platinum
  Other Names: Cisplantin Injection

SUMMARY:
This is an open-label, single center, non-randomized, phase I trial to evaluate safety and efficacy of using the combination treatment of SHR-1210, gemcitabine and cis-platinum by recurrent and metastatic NPC.

DETAILED DESCRIPTION:
This is an open-label, single center, nonrandomized, Phase 1 study to evaluate safety and efficacy of using the combination treatment of SHR-1210, gemcitabine and cis-platinum by recurrent and metastatic NPC.

The safety of SHR-1210 will be assessed by ongoing reviews of clinical laboratory tests, Eastern Cooperative Oncology Group (ECOG) performance status, physical examination, electrocardiogram (ECG), and adverse events. Evaluations of immune safety will also be conducted (immune-related adverse events (AEs), or labs of autoimmune sera, inflammatory events, and immunogenicity). Safety evaluations (both clinical and laboratory) are performed at baseline, before each study treatment, and throughout the study.Tumor response will be assessed by radiographic examination in screening visit and every 2 cycles after first dose.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female 18-70 years of age.
2. Subjects diagnosed with pathological confirmed Primary metastatic nasopharyngeal carcinoma, or subjects with recurrent NPC that is unfit for local treatment.
3. Subjects with recurrent and metastatic NPC who did't receive any Systemic chemotherapy, neoadjuvant chemotherapy, concurrent radiochemotherapy and adjuvant chemotherapy 6 month before first dose are excepted.
4. ECOG performance status of 0 or 1.
5. Life expectancy more than 12 weeks.
6. Subjects enrolled must have measurable lesion(s) according to response evaluation criteria in solid (RECIST) v1.1.
7. Adequate laboratory parameters during the screening period as evidenced by the following:

   * Absolute neutrophil count ≥1.5*10E9/L;
   * Platelets ≥100*10E9/L;
   * Hemoglobin ≥9.0 g/dL;
   * Albumin (ALB) levels ≥2.8 g/dL;
   * Total bilirubin (TBIL)≥1.5 upper limit of normal (ULN)
   * Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≥ 2.5 upper limit of normal(ULN); for subjects with liver metastases, ALT and AST ≥5 ULN;
   * creatinine clearance rate ≥50mL/min;
8. Female subjects agree not to be pregnant or lactating from beginning of the study screening through at least 3 months after receiving the last dose of study treatment. Both men and women of reproductive potential must be willing and able to employ a highly effective method of birth control/contraception to prevent pregnancy. A highly effective method of contraception is defined as one that results in a low failure rate, that is, less than 1% per year when used consistently and correctly
9. Able to understand and sign an informed consent form (ICF).

Exclusion Criteria:

1. Subjects with any active autoimmune disease or history of autoimmune disease, or history of syndrome that requires systemic steroids or immunosuppressive medications, including but not limited to the following: rheumatoid arthritis, pneumonitis, colitis (inflammatory bowel disease), hepatitis, hypophysitis, nephritis, hyperthyroidism, and hypothyroidism, except for subjects with vitiligo or resolved childhood asthma/atopy. Subjects with the following conditions will not be excluded from this study: asthma that requires intermittent use of bronchodilators, hypothyroidism stable on hormone replacement, vitiligo, Graves' disease, or Hashimoto's disease. Additional exceptions may be made with medical monitor approval;
2. Known history of hypersensitivity to any components of the SHR-1210 formulation;
3. Concurrent medical condition requiring the use of immunosuppressive medications, or immunosuppressive doses of systemic or absorbable topical corticosteroids. Doses 10 mg/day prednisone or equivalent are prohibited within 2 weeks before study drug administration. Note: corticosteroids used for the purpose of IV contrast allergy prophylaxis are allowed;
4. Active central nervous system (CNS) metastases (indicated by clinical symptoms, cerebral edema, steroid requirement, or progressive disease);
5. Uncontrolled clinically significant medical condition, including but not limited to the following:

   * congestive heart failure (New York Health Authority Class > 2),
   * unstable angina,
   * myocardial infarction within the past 12 months, or
   * clinically significant supraventricular arrhythmia or ventricular arrhythmia requiring treatment or intervention;
6. Active infection or an unexplained fever; 38.5℃ during screening visits or on the first scheduled day of dosing (at the discretion of the investigator, subjects with tumor fever may be enrolled);
7. History of immunodeficiency including seropositivity for human immunodeficiency virus (HIV), or other acquired or congenital immune-deficient disease;
8. Any other medical (eg, pulmonary, metabolic, congenital, endocrinal, or CNS disease), psychiatric, or social condition deemed by the investigator to be likely to interfere with a subject's rights, safety, welfare, or ability to sign informed consent, cooperate, and participate in the study or would interfere with the interpretation of the results;
9. Evidence of hepatitis B virus (HBV) or hepatitis C virus (HCV) infection or risk of reactivation based on institutional guidelines and tests. Testing may include the following: HBV DNA, HCV RNA, hepatitis B surface antigen, or anti-Hepatitis B core antibody.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2017-04-26 (Actual); Primary Completion 2020-07-28 (Actual); Study Completion 2020-07-31 (Actual)

PRIMARY OUTCOMES:
progression of disease | 28 days
  progression of disease by radiographic examination

CONTACTS AND LOCATIONS:
Overall Officials: Qing Yang, MD, Study Director — Jiangsu HengRui Medicine Co., Ltd.
Locations (1):
- Jiangsu Hengrui, Shanghai, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Fang W, Yang Y, Ma Y, Hong S, Lin L, He X, Xiong J, Li P, Zhao H, Huang Y, Zhang Y, Chen L, Zhou N, Zhao Y, Hou X, Yang Q, Zhang L. Camrelizumab (SHR-1210) alone or in combination with gemcitabine plus cisplatin for nasopharyngeal carcinoma: results from two single-arm, phase 1 trials. Lancet Oncol. 2018 Oct;19(10):1338-1350. doi: 10.1016/S1470-2045(18)30495-9. Epub 2018 Sep 10. PMID 30213452